CLINICAL TRIAL: NCT06890845
Title: Body Posture, Joint Range of Motion and Trunk Muscle Endurance in Relation to Low Back Pain in Tennis Players
Brief Title: Body Posture, Joint Mobility, and Trunk Muscle Endurance Related to Lower Back Pain in Tennis Players
Status: Completed | Type: Observational
Sponsor: Józef Piłsudski University of Physical Education (Other)
Responsible Party: Sponsor
Other Study IDs: Research#Group no 4
Record Dates: First submitted 2025-03-17; First posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2024-07

CONDITIONS: Low Back Pain
Keywords: low back pain, tennis, ROM, muscle endurance, posture
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Study Group (SG): Women and men amateur tennis players with LBP
- Comparison Group I (CGI): Women and men amateur tennis players without LBP
- Comparison Group II (CGII): Physically active women and men not engaged in asymmetric sports without LBP

SUMMARY:
The aim of this study was to determine the significance of the impact of external factors (self-evaluation of the subjects) and internal factors, including the range of motion in the spine and hip joints, trunk muscle endurance and body posture of tennis players, on the occurrence and severity of low back pain.

DETAILED DESCRIPTION:
The aim of the study was to compare tennis players with and without lower back pain (LBP) and individuals not engaged in asymmetric sports without LBP in terms of spinal flexion, extension, lateral bending range of motion, hip joint flexion, extension, internal and external rotation, modified seat and reach test results, trunk muscle endurance, body posture parameters, and survey information regarding training volume and stretching exercises. Identifying significant differences between participants with and without LBP could provide indications for modifying rehabilitation programs for amateur tennis players with LBP or for introducing preventive exercises targeting factors significantly influencing the occurrence of LBP in this population. Prior to the study, participants provided written consent and were informed of their right to withdraw from the study at any time.

ELIGIBILITY:
Inclusion Criteria:

* provided written consent to participate in the study

For Study Group:

* playing tennis at least 3 times per week for the past 2 years
* experiencing back pain in the last 6 months that prevented playing tennis

For Comprarison Group I:

* playing tennis at least 3 times per week for the past 2 years
* no lower back pain (confirmed via survey) in the last 6 months that would have prevented playing tennis

For Comparison Group II:

* no lower back pain (confirmed via survey)
* regular physical activity at least 3 times a week
* no participation in asymmetrical sports

Exclusion Criteria:

* lack of written consent to participate in the study,
* history of surgical procedures involving the spine or torso,
* severe musculoskeletal pathologies in the medical history, such as previous cancers in the torso area, vertebral fractures, structural scoliosis,
* inability to assume the required test positions.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants were recruited through announcements in tennis clubs, on internet portals, and on social media platforms within groups for amateur tennis players.
Sampling Method: Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Hip range of motion | Baseline
  The hip range of motion was measured using a digital inclinometer. During hip rotation measurement, the subject lay prone with the pelvis stabilized by a strap. The tested hip was in a neutral position with the knee flexed to 90 degrees. The inclinometer was zeroed along the tibial axis when the tibial plateau was parallel to the ground. The range of motion was the angular difference between the initial and final positions.
  For flexion, the subject lay supine with the non-tested lower limb stabilized. The inclinometer was zeroed parallel to the ground. The final position was where the thigh could no longer move further into flexion.
  For extension, the subject .lay supine with the pelvis at the edge of the table. The subject maximally flexed both hips. The subject held the non-tested lower limb with both hands. On the tested side, the lower limb hung freely off the table. The inclinometer was zeroed on a surface parallel to the ground, and in the final position of the test.
Spine range of motion | Baseline
  The measurement was conducted using a Baseline bubble inclinometer. For flexion, the patient stood in a relaxed position. The spinous processes of Th12 and S1 were palpated and marked. The inclinometer was zeroed at Th12, and the patient executed a full forward bend. The same was repeated at S1. The lumbar flexion range was the difference between readings at Th12 and S1.
  For extension, the patient also stood relaxed. Before measuring, the patient performed three maximum lumbar extensions. The inclinometer was zeroed at Th12, and the patient executed a maximum extension. The same procedure was repeated at S1. The lumbar extension range was the difference between readings at Th12 and S1.
  For lateral trunk flexion, the measurement was the distance between a point on the lateral thigh, where the tip of the third finger reached in a relaxed standing position, and a point on the thigh/shin after performing maximum lateral flexion.
Modified sit and reach test | Baseline
  To perform the test, the subject sat on the examination table in such a way that one lower limb rested on the floor with the knee flexed at 90 degrees, while the other limb was placed on the table with the knee joint extended. The subject positioned their hands in front of them, thumbs joined and palms facing down. With elbows fully extended, the subject reached as far forward as possible, placing their hands on the table. The distance from the tip of the third finger to the heel line was measured. Positive results indicated that the tip of the third finger extended beyond the heel line, while negative results indicated that it was positioned before the heel line.
Body posture | Baseline
  Posture assessment was conducted using the Diers Formetric 4D system, a non-invasive method with proven accuracy and reproducibility. This system employs surface topography for three-dimensional mapping of the subject's torso.
  The measurement followed the manufacturer's methodology. The subject stood 2 meters from the projector and camera, with foot placement marked on the treadmill. The back and neck were exposed, and undergarments adjusted to reveal the upper gluteal cleft. The subject assumed a relaxed standing position without posture correction. The examiner adjusted the projector height so that the central reference stripe aligned with the lower angle of the scapula. The device performed 12 scans in 6 seconds (2 Hz). The Diers software analyzed approximately 50,000 points on the subject's back, presenting a three-dimensional model of the spine with posture parameters.
Trunk muscle endurance | Baseline
  The protocol for assessing trunk muscle endurance was based on the McGill et al. (1999) method. [McGill, S. M., Childs, A., & Liebenson, C. (1999). Endurance times for low back stabilization exercises: Clinical targets for testing and training from a normal database. Archives of Physical Medicine and Rehabilitation, 80(8), 941-944. https://doi.org/10.1016/s0003-9993(99)90087-4]

SECONDARY OUTCOMES:
Oswestry Disability Index | Baseline
  The survey assessed the level of pain and disability associated with LBP.
Custom survey for individuals not playing tennis | Baseline
  The survey covered spinal pain, health status, physical activity, and the presence of chronic diseases
Custom survey for tennis players | Baseline
  The survey covered training volume, engagement in general conditioning and stretching exercises, presence of chronic diseases, history of injuries, and the level of spinal pain

CONTACTS AND LOCATIONS:
Locations (1):
- Mirai Clinic, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Avman MA, Osmotherly PG, Snodgrass S, Rivett DA. Is there an association between hip range of motion and nonspecific low back pain? A systematic review. Musculoskelet Sci Pract. 2019 Jul;42:38-51. doi: 10.1016/j.msksp.2019.03.002. Epub 2019 Mar 30. PMID 31030110
- [Background] Chun SW, Lim CY, Kim K, Hwang J, Chung SG. The relationships between low back pain and lumbar lordosis: a systematic review and meta-analysis. Spine J. 2017 Aug;17(8):1180-1191. doi: 10.1016/j.spinee.2017.04.034. Epub 2017 May 2. PMID 28476690